CLINICAL TRIAL: NCT03384992
Title: Targeted eHealth Intervention to Reduce Fear of Recurrence Among Breast Cancer Survivors: The FoRtitude Trial
Brief Title: Targeted eHealth Intervention to Reduce Fear of Recurrence Among Breast Cancer Survivors
Acronym: FoRtitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00036679; 1R21CA173193-01A1 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Fear of Cancer
Keywords: Fear of Cancer Recurrence; ehealth interventions; PROMIS; FoR
MeSH Terms: conditions — Breast Neoplasms; Pathophobia | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: FoRtitude includes three CSMs: (1) diaphragmatic breathing and relaxation, (2) cognitive restructuring, and (3) scheduled worry practice. The fourth intervention component is (4) telephone coaching. We assigned two levels (yes, no) to each component. Evaluating individual and combined intervention components, each with two levels, results in a classic full factorial design with 16 (2 x 2 x 2 x 2) experimental conditions
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Group 1 (Experimental): Participants were exposed to the following conditions: general health for week 1, diet-general information for week 2, and diet-BCSS information (breast cancer survivor-specific) for week 3. Telephone coaching was given.
  Interventions: Other: Telephone coaching; Other: Usual care
- Group 2 (Experimental): Participants were exposed to the one of the following usual care conditions: general health for week 1, diet-general information for week 2, and diet-BCSS information (breast cancer survivor-specific) for week 3.
  Interventions: Other: Usual care
- Group 3 (Experimental): Participants were exposed to the following conditions: cognitive restructuring for week 1, general health for week 2, and diet-general information and diet-BCSS information (breast cancer survivor-specific) for week 3. Telephone coaching was given.
  Interventions: Other: Cognitive restructuring; Other: Telephone coaching; Other: Usual care
- Group 4 (Experimental): Participants were exposed to the following conditions: cognitive restructuring for week 1, general health for week 2, and diet-general information and diet-BCSS information (breast cancer survivor-specific) for week 3.
  Interventions: Other: Cognitive restructuring; Other: Usual care
- Group 5 (Experimental): Participants were exposed to the following conditions: scheduled worry practice for week 1, general health for week 2, and diet-general information and diet-BCSS information (breast cancer survivor-specific) for week 3. Telephone coaching was given.
  Interventions: Other: Scheduled worry practice; Other: Telephone coaching; Other: Usual care
- Group 6 (Experimental): Participants were exposed to the following conditions: scheduled worry practice for week 1, general health for week 2, and diet-general information and diet-BCSS information (breast cancer survivor-specific) for week 3.
  Interventions: Other: Scheduled worry practice; Other: Usual care
- Group 7 (Experimental): Participants were exposed to the following conditions: cognitive restructuring for week 1, worry practice for week 2, and General Health and Diet (General and BCSS) for week 3. Telephone coaching was given.
  Interventions: Other: Cognitive restructuring; Other: Scheduled worry practice; Other: Telephone coaching; Other: Usual care
- Group 8 (Experimental): Participants were exposed to the following conditions: cognitive restructuring for week 1, scheduled worry practice for week 2, and General Health and Diet (General and BCSS) for week 3.
  Interventions: Other: Cognitive restructuring; Other: Scheduled worry practice; Other: Usual care
- Group 9 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, general health for week 2, and Diet - General and BCSS for week 3. Telephone coaching was given.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Telephone coaching; Other: Usual care
- Group 10 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, general health for week 2, and Diet - General and BCSS for week 3.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Usual care
- Group 11 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, cognitive restructuring for week 2, and General health and Diet (General and BCSS) for week 3. Telephone coaching was given.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Cognitive restructuring; Other: Telephone coaching; Other: Usual care
- Group 12 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, cognitive restructuring for week 2, and General health and Diet (General and BCSS) for week 3.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Cognitive restructuring; Other: Usual care
- Group 13 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, worry practice for week 2, and General health and Diet (General and BCSS) for week 3. Telephone coaching was given.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Scheduled worry practice; Other: Telephone coaching; Other: Usual care
- Group 14 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, scheduled worry practice for week 2, and General health and Diet (General and BCSS) for week 3.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Scheduled worry practice; Other: Usual care
- Group 15 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, worry practice for week 2, and cognitive restructuring for week 3. Telephone coaching was given.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Cognitive restructuring; Other: Scheduled worry practice; Other: Telephone coaching
- Group 16 (Experimental): Participants were exposed to the following conditions: Diaphragmatic breathing and relaxation for week 1, scheduled worry practice for week 2, and cognitive restructuring for week 3.
  Interventions: Other: Diaphragmatic breathing and relaxation; Other: Cognitive restructuring; Other: Scheduled worry practice

INTERVENTIONS:
Other: Diaphragmatic breathing and relaxation — Education on physiological effects of anxiety, instructions in diaphragmatic breathing and relaxation techniques, and audio-recordings 5-15 minutes in length that provide guided relaxation exercises (autogenic, imagery-based and progressive muscle relaxation).
  Arms: Group 10; Group 11; Group 12; Group 13; Group 14; Group 15; Group 16; Group 9
Other: Cognitive restructuring — Education on the thought-emotion connection and exercises designed to better understand cognitions associated with increased anxiety and tools to evaluate and replace anxiety-generating cognitions. Includes an interactive tool (thought record) participants complete to facilitate this process.
  Arms: Group 11; Group 12; Group 15; Group 16; Group 3; Group 4; Group 7; Group 8
Other: Scheduled worry practice — Education on the association between avoidance and increased anxiety, and instructions on actively thinking about feared events to reduce avoidance and engage healthy coping strategies. Interactive tool includes a video-based guided worry practice session and an interactive worksheet and timer.
  Arms: Group 13; Group 14; Group 15; Group 16; Group 5; Group 6; Group 7; Group 8
Other: Telephone coaching — BCS will receive 5 TeleCoaching calls over a period of 4 weeks, to include one introductory phone call, followed by 4 calls focused each week on the current CSM; if the participant is not randomized to a CSM, TeleCoaching will provide reflective listening and encouragement.
  Arms: Group 1; Group 11; Group 13; Group 15; Group 3; Group 5; Group 7; Group 9
Other: Usual care — Includes general health, diet-general information and diet-BCSS (breast cancer survivor-specific) information.
  Arms: Group 1; Group 10; Group 11; Group 12; Group 13; Group 14; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7; Group 8; Group 9

SUMMARY:
The FoRtitude trial aims to evaluate an eHealth intervention designed to teach breast cancer survivors strategies to manage anxiety about cancer recurrence. The eHealth intervention includes educational content and interactive tools, designed to teach coping strategies and/or inert content, depending on the study participant's randomization assignment. The FoRtitude study will examine whether three coping strategies (relaxation training, cognitive restructuring, worry practice) are more effective than general health-related content in reducing fear of cancer recurrence.

DETAILED DESCRIPTION:
The purpose of the FoRtitude trial is to develop and evaluate a targeted eHealth intervention designed to teach breast cancer survivors (BCS) coping strategies to manage fear about cancer recurrence (FoR). FoRtitude, a web-based program with interactive text messaging capabilities, was created to deliver a targeted intervention for BCS with moderate to severe FoR. FoRtitude consists of didactic content presented in written and video-based formats and interactive tools, designed to teach coping strategies. Commonly used cognitive behavior therapy (CBT) techniques were tailored to the management of FoR and included diaphragmatic breathing and relaxation, cognitive restructuring, and scheduled worry practice. Participants are encouraged to use the FoRtitude site several times per week over a period of 4 weeks. The investigators employed principles of user-centered design to create the FoRtitude website and incorporated feedback from 17 BCS to refine site content and improve FoRtitude usability.

After refining the FoRtitude site, the investigators will conduct a randomized controlled trial using the Multiphase Optimization Strategy (MOST) to individually evaluate three coping strategies; each coping strategy will be compared to health management content. Inert content includes general health information and managing comorbid illnesses, information on general nutrition, and information on nutritional topics of interest to BCS. Half of the participants will be randomized to receive telecoaching, which included 3-4 telephone-based brief sessions with a motivational interviewer, aimed at improving adherence to use of the FoRtitude site. Participants will complete questionnaires at baseline, 4 weeks (immediately after completing the FoRtitude site) and at 8 weeks.

Study hypotheses:

1. BCS randomized to Relaxation training will report a greater reduction in fear of cancer recurrence from pre-post intervention than BCS randomized to inert (health management) content
2. BCS randomized to Cognitive restructuring will report a greater reduction in fear of cancer recurrence from pre-post intervention than BCS randomized to inert (health management) content
3. BCS randomized to Scheduled Worry practice will report a greater reduction in fear of cancer recurrence from pre-post intervention than BCS randomized to inert (health management) content
4. BCS randomized to receive Telecoaching will demonstrate higher adherence to using the FoRtitude site and will report a greater reduction in fear of cancer recurrence from pre-post intervention compared to BCS randomized to no Telecoaching
5. BCS randomized to a higher number of coping strategies will report a greater reduction in fear of cancer recurrence from pre-post intervention than BCS randomized to receive all inert content or fewer coping strategies (dose-response effect)

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of breast cancer, non-metastatic, stage I-III
* Completed primary treatment for breast cancer (surgery, chemotherapy and/or radiation therapy, current hormonal treatment allowable)
* No current evidence of disease

  1. Greater than 1 year post treatment (for phase I interviews and usability testing)
  2. Between 1 and 10 years post-treatment (for Phase I field testing and Phase II)
* Good overall functional status as evidenced by ECOG Performance Status < 3
* At least 18 years of age (for Phase I only)
* At least 19 years of age (for Phase 2 only)
* Able to speak and read English
* Able to provide informed consent
* Clinically significant FoR, measured by the 9-item FCRI severity scale using established cut-off

  a. Patients may be eligible for Phase I and Phase IV of the study regardless of their FCRI score
* Cellular telephone with SMS messaging capability and access to a computer with broadband Internet access
* Self-reported familiarity with the Internet per Internet Usage Patterns Measure
* For Phase III, participants must have participated in Phase II
* For Phase IV, participants must be a self-identified African American breast cancer survivor that is willing to review site content and provide feedback in addition to meeting inclusion criteria above (with exception of FCRI severity scale score)

Exclusion Criteria:

* Visual, hearing, voice, or motor impairment that would prevent completion of study procedures
* Diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, or other diagnosis for which participation in this trial is either inappropriate or dangerous
* Hazardous substance or alcohol use
* Suicidal ideation, plan, intent
* Dementia
* Or if the participant is deemed ineligible by the investigators for reasons not otherwise specified.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-12-05 (Actual); Study Completion 2015-12-05 (Actual)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory (FCRI) total score (minus Coping and Reassurance subscales) | Baseline to Week 8 change score
  Questionnaire aims to better understand the experience of worries about cancer recurrence. Scaled from 1-4 with 4 being "all the time" and 1 being "never". The FCRI is the only FoR measure validated using interview to define 'caseness' and has demonstrated reliability and validity with English speaking survivors. FCRI total score to be calculated without including the Coping and Reassurance subscales defined a priori and determined by FoR theoretical model.

SECONDARY OUTCOMES:
Impact of Events Scale - Revised | Baseline to Week 8 change score
  Questionnaire to assess illness-related distress and post-truamatic type anxiety
Concerns about Recurrence Scale (CARS) - 4 item severity score | Baseline to Week 8 change score
  Questionnaire to assess concerns about recurrence among BCS
PROMIS Anxiety Computer adaptive test | Baseline to Week 8 change score
  Questions administered using a computer adaptive test-based algorithm to assess overall anxiety
PROMIS Depression Computer adaptive test | Baseline to Week 8 change score
  Questions administered using a computer adaptive test-based algorithm to assess depression
PROMIS Sleep Disturbance Computer adaptive test | Baseline to Week 8 change score
  Questions administered using a computer adaptive test-based algorithm to assess sleep disturbances
PROMIS Fatigue Computer adaptive test | Baseline to Week 8 change score
  Questions administered using a computer adaptive test-based algorithm to assess fatigue
PROMIS Global Health | Baseline to Week 8 change score
  Questionnaire to assess overall health and health-related quality of life
PROMIS Applied Cognition Computer adaptive test | Baseline to Week 8 change score
  Questions administered using a computer adaptive test-based algorithm to assess patient-reported cognitive impairments
Breast Cancer Self-Efficacy scale (BCSE) | Baseline to Week 8 change score
  Questionnaire to assess confidence in one's ability to manage breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Wagner, Ph.D., Principal Investigator — Wake Forest University Health Sciences

REFERENCES:
- [Derived] Beeler DM, Jeter E, Leitzelar BN, Price SN, Hall DL, Raper PJ, Levine BJ, Dunsmore VJ, Tooze JA, Duffecy J, Victorson D, Gradishar W, Saphner T, Smith ML, Penedo F, Mohr DC, Cella D, Wagner LI. A qualitative examination of cognitive behavioral therapy strategies and health management content to reduce fear of cancer recurrence among breast cancer survivors: Results from the FoRtitude study. J Health Psychol. 2025 Jul 28:13591053251354867. doi: 10.1177/13591053251354867. Online ahead of print. PMID 40721359
- [Derived] Lucas AR, Pan JH, Ip EH, Hall DL, Tooze JA, Levine B, Mohr DC, Penedo FJ, Cella D, Wagner LI. Validation of the Lee-Jones theoretical model of fear of cancer recurrence among breast cancer survivors using a structural equation modeling approach. Psychooncology. 2023 Feb;32(2):256-265. doi: 10.1002/pon.6076. Epub 2023 Jan 9. PMID 36468339